CLINICAL TRIAL: NCT05492344
Title: Personalized Mechanical Ventilation Guided by UltraSound in Patients With Acute Respiratory Distress Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PEGASUS
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: ARDS, Human; Lung Ultrasound; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized ventilation (Experimental): If a patient is assigned to the intervention group, ventilator settings will be adjusted based on the lung morphology (focal or non focal) results of the lung ultrasound.
  Interventions: Other: Personalized ventilation
- Standard care (Active Comparator): Patients assigned to the control group will be ventilated according to the current standard of care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Personalized ventilation — Patients who are randomized for personalized ventilation with FOCAL ARDS will receive the following ventilator settings:
  * Positive end-expiratory pressure (PEEP) ≤ 9 cm water (H2O)
  * Tidal volume: 6 to 8 mL/kg predicted body weight (PBW)
  * Daily prone positioning
  LUS will be repeated every 48-72 hours in supine position for the focal ARDS patients to assess whether they have developed non-focal ARDS during admission. In that case, patients will from then on be treated according non-focal personalized treatment protocol.
  Patients who are randomized for personalized ventilation with Non-FOCAL ARDS will receive the following ventilator settings:
  * PEEP ≥ 15 cm H2O
  * Tidal volume: 4 to 6 mL/kg PBW
  * Daily recruitment maneuver
  Arms: Personalized ventilation
Other: Standard care — Patient who are randomized in the control group will receive standard care
  * Tidal volume: 6 mL/kg PBW
  * PEEP and FiO2 according to the low PEEP and high fraction of inspired oxygen (FiO2) table of the AlVEOLI study
  * Prone positioning if the Partial Pressure of Oxygen (PaO2) /FiO2 ratio is < 150 mmHg
  Arms: Standard care

SUMMARY:
Rationale Acute respiratory distress syndrome (ARDS) is a frequent cause of hypoxemic respiratory failure with a mortality rate of approximately 30%. The identification of ARDS phenotypes, based on focal or non-focal lung morphology, can be helpful to better target mechanical ventilation strategies of individual patients. Lung ultrasound (LUS) is a non-invasive tool that can accurately distinguish 'focal' from 'non-focal' lung morphology. The investigators hypothesize that LUS-guided personalized mechanical ventilation in ARDS patients will lead to a reduction in 90-day mortality compared to conventional mechanical ventilation.

DETAILED DESCRIPTION:
Objective The aim of this study is to determine if personalized mechanical ventilation based on lung morphology assessed by LUS leads to a reduced mortality compared to conventional mechanical ventilation in ARDS patients.

Study design The PEGASUS study is an investigator-initiated multicenter randomized clinical trial (RCT) with a predefined feasibility and safety evaluation after a pilot phase.

Study population This study will include 538 consecutively admitted invasively ventilated adult intensive care unit (ICU) patients with moderate or severe ARDS. There will be a predefined feasibility and safety evaluation after inclusion of the first 80 patients.

Intervention Patients will receive a LUS exam within 12 hours after diagnosis of ARDS to classify lung morphology as focal or non-focal ARDS. Immediately after the LUS exam patients will be randomly assigned to the intervention group, with personalized mechanical ventilation, or the control group, in which patients will receive standard care.

Main study parameters/endpoints The primary endpoint is all cause mortality at day 90 (diagnosis of ARDS considered as day 0). Secondary outcomes are mortality at 28 days, ventilator free days (VFD) at day 28, ICU length of stay, ICU mortality, hospital length of stay, hospital mortality and number of complications (VAP, pneumothorax and need for rescue therapy). After a pilot phase, feasibility of LUS, correct interpretation of LUS images and correct application of the intervention within the safe limits of mechanical ventilation is evaluated to inform a stop-go decision.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Patient burden and risks are low as the ventilation methods in this study are already commonly used in ICU practice; the collection of general data from hospital charts and (electronic) medical records systems causes no harm to the patients; LUS is not uncomfortable.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a participating ICU,
* invasively ventilated and
* fulfil the Berlin criteria for moderate or severe ARDS.

Exclusion Criteria:

* Age under 18,
* participation in other interventional studies with conflicting endpoints,
* conditions in which LUS is not feasible or possible (e.g. subcutaneous emphysema, morbid obesity or wounds),
* mechanical ventilation for longer than 7 consecutive days in the past 30 days,
* history of ARDS in the previous month,
* body-mass index higher than 40 kg/m²,
* intracranial hypertension,
* broncho-pleural fistula,
* chronic respiratory diseases requiring long-term oxygen therapy or respiratory support,
* pulmonary fibrosis with a vital capacity < 50% (severe or very severe),
* previously randomized in the PEGASUS study
* ECMO
* patients who are moribund or facing end of life and
* no informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 90 days after inclusion
  Any death during ICU- or hospital-stay at day 90

SECONDARY OUTCOMES:
All-cause mortality | 28 days after inclusion
  Any death during ICU- or hospital-stay at day 28
Ventilator free days | 28 days after inclusion
  Duration of ventilation in survivors
ICU length of stay | 90 days after inclusion
  Length of stay in the intensive care unit
ICU mortality | 90 days after inclusion
  Mortality in the ICU
Hospital length of stay | 90 days after inclusion
  Length of stay in the hospital
Hospital mortality | 90 days after inclusion
  Mortality in the hospital
Number of patients with Complications | 90 days after inclusion
  Ventilator associated pneumonia and pneumothorax
Number of patients with Adjunctive therapies | 90 days after inclusion
  Extracorporeal membrane oxygenation (ECMO), recruitment, prone position
Number of patients with Rescue therapies | 90 days after inclusion
  Inhaled vasodilators, airway pressure release ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Lieuwe DJ Bos, Dr., Principal Investigator — Amsterdam UMC, location AMC
Locations (10):
- Chu-Brugmann, Brussels, Belgium
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Nordsjaellands Hospital, Hillerød
- Evaggelismos Hospital, Athens, Greece
- Galway University Hospitals, Galway, Ireland
- Italy (2):
  - Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti, Bari
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
- Netherlands (2):
  - Amsterdam UMC, location VUmc, Amsterdam, North Holland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
- Centralny Szpital Kliniczny MSWiA, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sinnige JS, Smit MR, Alam MJ, Chowdhury MNH, Costa V, de Castro HSMB, Daszuta D, Filippini DFL, Ghose A, de Grooth HJ, Hein L, Hermans G, Hildebrandt T, Itenov TS, Ischaki E, Klompmaker P, Laffey J, McMahon A, McNicholas B, Mousa A, Paulus F, Pedersen UG, Pellegrini M, Pezzuto M, Povoa P, Pierrakos C, Pisani L, Roca O, Schultz MJ, Spadaro S, Szuldrzynski K, Theodorou E, Tuinman PR, Wamberg CA, Zimatore C, Bos LDJ; PEGASUS investigators. Personalized mechanical ventilation guided by lung ultrasound in patients with ARDS: a pilot phase of a randomized clinical trial. Intensive Care Med Exp. 2025 Dec 22;13(1):135. doi: 10.1186/s40635-025-00835-8. PMID 41423518
- [Derived] Sinnige JS, Smit MR, Ghose A, de Grooth HJ, Itenov TS, Ischaki E, Laffey J, Paulus F, Povoa P, Pierrakos C, Pisani L, Roca O, Schultz MJ, Szuldrzynski K, Tuinman PR, Zimatore C, Bos LDJ; PEGASUS investigators. Personalized mechanical ventilation guided by ultrasound in patients with acute respiratory distress syndrome (PEGASUS): study protocol for an international randomized clinical trial. Trials. 2024 May 7;25(1):308. doi: 10.1186/s13063-024-08140-7. PMID 38715118